CLINICAL TRIAL: NCT03828773
Title: PTX3 Genetically Stratified Randomized Double-blinded Allocation Event-driven Clinical Trial for Antifungal Prophylaxis in Patients With Acute Myeloid Leukemia
Brief Title: PTX3-targeted Antifungal Prophylaxis
Acronym: PTX3AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bochud Pierre-Yves (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Bochud Pierre-Yves, Associate Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-01671
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Candidiasis; Fungal Infection; Acute Myeloid Leukemia; Genetic Predisposition; Aspergillosis
MeSH Terms: conditions — Candidiasis; Mycoses; Leukemia, Myeloid, Acute; Genetic Predisposition to Disease; Aspergillosis | interventions — posaconazole; Fluconazole

STUDY DESIGN:
Intervention Model Description: prospective genetically-stratified randomized double-blind event-driven multicentre clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational medicinal products will be known by all roles but the arm allocation based on a genetic analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-risk PTX3 SNPs (Other): risk predicted by genotyping two PTX3 single nucleotide polymorphisms (SNPs): homozygous for rs230561 and/or rs381652
  Interventions: Drug: Posaconazole; Drug: Fluconazole
- low-risk PTX3 SNPs (Other): risk predicted by genotyping two PTX3 single nucleotide polymorphisms (SNPs): other than homozygous for rs230561 and/or rs381652
  Interventions: Drug: Posaconazole; Drug: Fluconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole is a triazole with broad-spectrum activity, to include Candida species, Aspergillus species, and other fungal pathogens, including the Zygomycetes. Posaconazole is available as slow release tablets (300mg/day) and as intravenous (IV) formulation (300mg/day) and is licensed and approved in Switzerland for the prevention of IFI, including mold and yeast infections, in patients >18 years who are at high risk of developing these types of infection (patients with long-term neutropenia or HCT recipients). Furthermore, international guidelines recommend posaconazole for primary antifungal prophylaxis in high-risk patients, such as AML patients with prolonged neutropenia. Posaconazole is available in Switzerland under the name of Noxafil® in capsules of 100mg, suspension of 40mg/mL and intravenous formulation of 300mg/16.7 mL.
  Other Names: Noxafil
Drug: Fluconazole — Fluconazole is an antifungal with activity against most Candida species. Fluconazole is licensed and approved in Switzerland for prophylaxis of IC in patients with neutropenia induced by chemotherapy or radiotherapy at a daily dose of 200 to 400 mg once daily. Fluconazole (200 mg or 400 mg once daily) is still currently used as primary antifungal prophylaxis (standard of care) in all 7 centers participating in this trial. Fluconazole is available in Switzerland under the name of Diflucan® in capsules of 50 mg, 150 mg and 200 mg and in powder for preparation of suspension (50 mg/5 ml and 200 mg/5 ml (forte)) or perfusion (2 mg/1 ml). Several generics of Diflucan® are authorized in Switzerland. Prescribing Diflucan® or any of its generics will remain at the discretion of and based on the standard operating procedures (SOP) at each institution.
  Other Names: Diflucan

SUMMARY:
This is a prospective genetically-stratified randomized double-blind event-driven multicentre clinical trial to assess the efficacy of posaconazole-based antifungal prophylaxis allocation strategies for patients with acute myeloid leukemia who receive induction chemotherapy. Allocation strategy based on an invasive mold infection genetic risk will be double-blinded.

DETAILED DESCRIPTION:
Background:

Invasive mold infections (IMI, grouping infections due to Aspergillus spp [IA] and non-Aspergillus mold) are a major concern in hematological patients, such as those with acute myeloid leukemia (AML) or myelodysplastic syndrome in transformation (MDSit), collectively named AML/MDSit in this protocol, or those undergoing hematopoietic cell transplantation (HCT), with incidence and mortality rates ranging between 3-15% and 25-45%, respectively. Primary antifungal prophylaxis has become the standard of care in such patients. Historically, fluconazole (inactive against IA) was used as prophylaxis and allowed for significant decrease in invasive candidiasis (IC). More recently, posaconazole (a broad-spectrum azole active against IA and other non-Aspergillus filamentous molds) was approved for primary antifungal prophylaxis in high-risk patient categories. However, universal prophylaxis with posaconazole has been challenged, based on the relatively low incidence of IMI and the large number of patients needed to treat. Moreover, administration of broad-spectrum azoles is costly and associated with a large number of complications. Hence, there is an urgent need to optimize antifungal prophylaxis by identifying those patients with the highest risk for IMI to receive a broad-spectrum azole. Pentraxin-3 (PTX3), a pattern recognition receptor, recognizes and binds to Aspergillus conidia, facilitates opsonization and subsequently leads to complement and phagocyte activation. Two single nucleotide polymorphisms (SNPs) in the gene encoding PTX3 have been identified as strong predictors for IA and/or IMI in human studies. What makes PTX3 SNPs different and important in clinical practice is: (i) the extent and reproducibility of basic science data with regards to PTX3 and IA, (ii) the validation of PTX3 SNPs associations with IA in many different patient populations, and (iii) the high frequency of minor allele in the general population. The investigators hypothesize that PTX3 SNPs could be used to identify patients at high risk for IMI, who will benefit the most from antifungal prophylaxis with broad-spectrum azoles.

Overall objective:

The overall aim of this project is to assess the effectiveness of the use of posaconazole-based antifungal prophylaxis in AML/MDSit patients in high risk group (single or double single homozygotes PTX-3 SNPs). Exploratory objectives are to assess the effectiveness of PTX3 SNPs testing to stratify the use of posaconazole-based antifungal prophylaxis in AML/MDSit patients according to low or high risk genotypes.

Methods:

Eligible patients will be tested by competitive allele-specific Polymerase Chain Reaction (PCR) from blood-extracted DNA samples for the presence of PTX3 SNPs rs230561 and rs3816527. Randomisation based on genetic testing will be performed at the latest 24h after the first neutropenia day (D0). Patients will be stratified based on genotyping results in two unbalanced strata: stratum A (high-risk PTX3 SNPs) to be randomized 1:1 posaconazole prophylaxis vs fluconazole and stratum-B (low-risk PTX3 SNPs) to be randomized 1:3 in favour of Fluconazole. Patients will be assessed for a diagnosis of possible, probable or proven Invasive Fungal Infections (IFI) based on consensus definition guidelines by the European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC/MSG) groups during 180 days after prophylaxis initiation.

Impact:

The results of this study may contribute to the optimization of primary antifungal prophylaxis, by preventing IMI while limiting the use of broad-spectrum azoles, thus decreasing complications and costs. This study is one of the first interventional clinical trials to use genetic factors for risk stratification in the field of hematology and infectious diseases, a concept frequently emphasized, however barely transcribed in practice, as precision medicine. Furthermore, the scope of the proposed study expands beyond the specific patient population. The results of this study could be used in the design and initiation of similar efforts in other high-risk patient categories, including allogeneic HCT and solid organ transplant (SOT) recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent according to national/local regulations.
2. Age ≥18 years.
3. Diagnosis of Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome in transformation (MDSit) treated with an intensive chemotherapy regimen, including induction / consolidation / salvage remission chemotherapy.
4. Planned hospital admission for the duration of the neutropenic phase (absolute neutrophils count <500 cells/mm3).

Exclusion Criteria:

1. Patients with neutropenia (absolute neutrophils count<500 cells/mm3) upon presentation and prior to chemotherapy initiation.
2. Patients with a diagnosis of acute promyelocytic leukemia (APL) or AML-M3.
3. Patients with known history of allergy, hypersensitivity or serious reaction to azole antifungals
4. Women who are pregnant (positive blood/urine pregnancy test within 10 days before randomization) or breast-feeding.
5. Diagnosis and treatment for an Invasive Fungal Infection (IFI) within 3 months prior to study enrolment and an Invasive Mold Infection (IMI) at any point prior to or at the time of enrolment.
6. Severe liver dysfunction, defined as at least one of the following markers: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) or alkaline phosphatase above >5x upper limit of normality: and/or total bilirubin above >3x upper limit of normality.
7. Patients with an ECG with a prolonged QTc interval: QTc greater than 450 msec for men and greater than 470 msec for women.
8. Patients who are receiving and cannot discontinue the following drugs at least 24 hours prior to randomization: terfenadine, astemizole, cisapride, pimozide, halofantrine or quinidine (because of the possibility of QT prolongation), sirolimus, rifampin, rifabutin, carbamazepine, long-acting barbiturates (e.g., phenobarbital, mephobarbital), ritonavir, efavirenz, or ergot alkaloids (e.g., ergotamine, dihydroergotamine).
9. Serious uncontrolled concomitant disease or comorbidity that, in the opinion of the investigator, may compromise adherence to the study protocol.
10. Receipt of a prior allogeneic Hematopoietic Cell Transplantation (HCT).
11. Previous exposure to mold-active prophylaxis (>48 hours within 7 days of inclusion).
12. Patients with relapsed leukemia already included in the trial.
13. Patient not affiliated to the French social security system
14. Patient under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of proven and probable invasive mold infection (IMI) | Day 180
  The cumulative incidence of proven and probable invasive mold infection (IMI) (based on published consensus guidelines by the EORTC/MSG groups and after validation by an independent adjudication committee of infectious disease experts blinded to treatment arms) in the intention-to-treat (ITT) population by day 180.

SECONDARY OUTCOMES:
Cumulative incidence of possible invasive mold infection (IMI) | Day 180
  The cumulative incidence of possible invasive mold infection (IMI) (based on published consensus guidelines by the EORTC/MSG groups and after validation by an independent adjudication committee of infectious disease experts blinded to treatment arms) by day 180 in the ITT population.
Cumulative incidence of probable and proven Invasive Fungal Infections (IFI) | Day 180
  The cumulative incidence of probable and proven Invasive Fungal Infections (IFI) (based on published consensus guidelines by the EORTC/MSG groups and after validation by an independent adjudication committee of infectious disease experts blinded to treatment arms), namely: (a) all IFI, (b) Invasive Aspergillosis (IA) only and (c) Invasive Candidiasis (IC) only in the ITT patient population by day 180.
Time to probable and proven invasive mold infection (IMI) | Day 180
  The time to probable and proven invasive mold infection (IMI) (based on published consensus guidelines by the EORTC/MSG groups and after validation by an independent adjudication committee of infectious disease experts blinded to treatment arms) during 180 days in the ITT population
Cumulative incidence of mortality | Day 180
  The cumulative incidence of mortality in the ITT population by day 180.
Time to first use and number of patient-days of amphotericin B/echinocandin | Day 180
  The time to use of amphotericin B/echinocandin in the ITT population during 180 days.
Frequency/distribution of adverse events (AE) of interest | Day 180
  The frequency/distribution of AE of interest in posaconazole and fluconazole treated participants in the ITT population during 180 days, namely:
  1. Hepatotoxicity, defined by elevation of at least one of the following markers above >5x upper limit of normal: transaminases, alkaline phosphatase and/or above >3x upper limit of normal total bilirubin
  2. New QTc prolongation, defined as QTc >450 msec for men and >470 msec for women
Treatment success versus failure | Day 180
  Treatment failure was defined as any of the following: proven or probable IFI, administration of any other systemically administered antifungal treatment for more than 10 consecutive days, discontinuation of prophylaxis for any other reason (e.g. severe adverse event associated with the study medication), death, loss to follow-up, or withdrawal from the study.
Cumulative incidence of probable and proven invasive fungal infections (IFI) in per protocol population | Day 180
  The cumulative incidence of probable and proven invasive fungal infections (IFI) (based on published consensus guidelines by the EORTC/MSG groups and after validation by an independent adjudication committee of infectious disease experts blinded to treatment arms) , namely: all Invasive Fungal Infections (IFI), all Invasive Mold Infections (IMI), Invasive Aspergillosis (IA) only and Invasive Candidiasis (IC) only in the per protocol (PP) population by day 180.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Bochud, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (9):
- Belgium (3):
  - Ghent University Hospital, Ghent, Belgium
  - AZ Sint-Jan Hospital, Bruges
  - University Hospital Leuven (UZ Leuven), Leuven
- Henri Mondor Hospital, Créteil, Île-de-France Region, France
- Switzerland (5):
  - Cantonal Hospital Aarau, Aarau, Aarau
  - University Hospital Basel, Basel, Basel
  - Cantonal Hospital HFR, Fribourg, Canton of Fribourg
  - University Hospital of Geneva (HUG), Geneva, Canton of Geneva
  - University Hospital of Lausanne / Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud